CLINICAL TRIAL: NCT01213446
Title: A Phase III Open-label, Multi-centre Study to Assess the Pharmacokinetics, Efficacy, and Safety of Biostate® in Paediatric Subjects With Von Willebrand Disease
Brief Title: Study of Biostate® in Children With Von Willebrand Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-BIO-08-52; 2009-017753-34 (EudraCT Number); 1494 (Other: CSL Behring)
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Von Willebrand Disease
Keywords: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biostate (Experimental)
  Interventions: Biological: Biostate

INTERVENTIONS:
Biological: Biostate — PK component: Single bolus infusion of 80 IU VWF:RCo/kg administered intravenously on Day 1, and approximately Day 180 in Type 3 VWD subjects only.
  Efficacy component: Repeated bolus doses over 12 months as required to manage VWD condition.

SUMMARY:
This is an open-label study to investigate the pharmacokinetics (PK), efficacy, and safety of a von Willebrand Factor/Factor VIII (VWF/FVIII), Biostate, in children with Von Willebrand disease (VWD) in whom treatment with a VWF product is required for prophylactic therapy, haemostatic control during surgery, or control of a non-surgical, spontaneous, or traumatic bleeding event.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 0 and <12 years of age
* Diagnosed with VWD Type 1, 2A, or 3
* Desmopressin acetate (DDAVP) treatment is ineffective, contraindicated, or not available for subject
* von Willebrand factor: ristocetin cofactor (VWF:RCo) is <20% at screening or the subject has a history of VWF:RCo <10%
* Evidence of vaccination against hepatitis A and B or presence of antibodies against hepatitis A and B due to either a previous infection or prior immunization
* Written informed consent given

Exclusion Criteria:

* Active bleeding immediately prior to initial PK period
* Received treatment with DDAVP or a VWF concentrate product for their VWD in the 5 days prior to their first study treatment
* Have received aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs) within 7 days of commencing the PK period.
* Known history or suspicion of having VWF or FVIII inhibitors
* Acute or chronic medical condition, other than VWD, which may affect the conduct of the study
* Known or suspected hypersensitivity or previous evidence of severe side effects to other FVIII/VWF concentrates
* Participation in a clinical study or use of an investigational compound in another study in the 3 months preceding study start
* Unwillingness and/or inability to comply with the study requirements

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Haemostatic efficacy | From Day 1 until final study visit
Incremental Recovery of VWF | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1 and 6 months after initial dose
Incremental Recovery of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Half-life of VWF | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1 and 6 months after initial dose
Half-life of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Area under the concentration curve (AUC) of VWF | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1 and 6 months after initial dose
AUC of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Maximum plasma concentration (Cmax) of VWF | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1 and 6 months after initial dose
Maximum plasma concentration (Cmax) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Minimum plasma concentration (Cmin) of VWF | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1 and 6 months after initial dose
Minimum plasma concentration (Cmin) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Time to maximum concentration (tmax) of VWF | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1 and 6 months after initial dose
Time to maximum concentration (tmax) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Mean residence time (MRT) of VWF | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1 and 6 months after initial dose
Mean residence time (MRT) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Clearance (CL) of VWF | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1 and 6 months after initial dose
Clearance (CL) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1
Volume of distribution of steady state (Vss) of VWF | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1 and 6 months after initial dose
Volume of distribution of steady state (Vss) of FVIII | Samples taken prior and then 0.5, 4, 8, 24, and 48 h after the infusion on Day 1

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) per infusion | 13 months
Severity of AEs per infusion | 13 months
Severity of AEs per subject | 13 months
Relatedness of AEs per infusion | 13 months
Relatedness of AEs per subject | 13 months
Development of VWF inhibitors | Sample taken at baseline, then every 3 months up to 12 months
Development of FVIII inhibitors | Sample taken at baseline, then every 3 months up to 12 months
Frequency of adverse events (AEs) per subject | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (7):
- Belarus (2):
  - Study site, Homyel
  - Study site, Minsk
- Study site, Tbilisi, Georgia
- Study site, Bremen, Germany
- Study site, Guatemala City, CP, Guatemala
- Study site, Beirut, Lebanon
- Study Site, Lviv, Ukraine